CLINICAL TRIAL: NCT01194219
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Efficacy and Safety Study of Apremilast (CC-10004) in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Study to Evaluate Safety and Effectiveness of Oral Apremilast (CC-10004) in Patients With Moderate to Severe Plaque Psoriasis
Acronym: ESTEEM 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSOR-008
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2020-04

CONDITIONS: Plaque Psoriasis
Keywords: Plaque Psoriasis
MeSH Terms: interventions — apremilast; Therapeutics; Phototherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Apremilast (Active Comparator): Subjects initially randomized to apremilast 30 mg twice a day, and who demonstrate a PASI 75 response at Week 32 will be randomized (1 to 1) to either continue to receive apremilast 30 mg ) BID or to receive placebo (until effect is lost). At the time effect is lost, subjects will be treated with apremilast 30 mg twice a day for the duration of their participation in the study.
  Interventions: Drug: Apremilast; Drug: Placebo
- Placebo (Placebo Comparator): Subjects initially randomized to placebo, are assigned to apremilast 30 mg twice a day beginning at Week 16 for the duration of the subject's participation in the study.
  Interventions: Drug: Apremilast; Drug: Placebo
- Apremilast 30 mg (Active Comparator): Apremilast 30 mg by mouth (PO) twice a day (BID). Participants initially randomized to apremilast 30 mg BID, and who were able to demonstrate a Psoriasis Area Severity Index (PASI) -75 response at week 32 were randomized (1 to 1) to either apremilast 30 mg BID or oral placebo (until effect is lost). At relapse/loss of response to therapy prior to Week 52 (the time at which 75% improvement in PASI score compared to baseline was lost) or at Week 52, participants were re-treated with apremilast 30 mg BID for the duration of their participation in the study. Non-responders or partial responders (PASI response <75) received additional topical therapies or phototherapy beginning at Week 32.
  Interventions: Drug: Apremilast; Drug: Placebo; Drug: Topical treatments or phototherapy

INTERVENTIONS:
Drug: Apremilast
  Other Names: CC-10004; Otezla
Drug: Placebo — Identical matching placebo
Drug: Topical treatments or phototherapy — At week 32, participants considered partial responders or non-responders had the option of adding topical therapies and/or phototherapy to their treatment regimen.
  Other Names: Corticosteroid creams; Light Therapy
  Arms: Apremilast 30 mg

SUMMARY:
This study evaluated the effects of an called apremilast. Apremilast works by lowering some of the chemicals that affect psoriasis and therefore improves the symptoms of psoriasis. The purpose of this study was to test apremilast and compare its effects to placebo (an inactive substance which contains no medicine but is in the same form as the drug). This study was able to test for efficacy (improvement of signs and symptoms) and safety of apremilast in patients with moderate to severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, ≥ 18 years of age at the time of signing the informed consent document
2. Diagnosis of chronic plaque psoriasis for at least 12 months prior to Screening

   a. Have moderate to severe plaque psoriasis at Screening and Baseline
3. Must meet all laboratory criteria
4. Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. FCBP who engage in activity in which conception is possible must use 2 forms of contraception as described by the Study Doctor while on study medication and for at least 28 days after taking the last dose of study medication
5. Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (latex condom or any nonlatex condom NOT made out of natural [animal] membrane [eg, polyurethane]) while on study medication and for a least 28 days after the last dose of study medication.

Exclusion Criteria:

1. Other than psoriasis, history of any clinically significant (as determined by the Investigator) or other major uncontrolled disease.

   .
2. Pregnant or breast feeding
3. History of allergy to any component of the study drug
4. Hepatitis B surface antigen positive at Screening
5. Anti-hepatitis C antibody positive at Screening
6. Active tuberculosis (TB) or a history of incompletely treated TB
7. Clinically significant abnormality on 12-Lead Electrocardiogram (ECG) at Screening
8. Clinically significant abnormal chest x-ray
9. History of positive human immunodeficiency virus (HIV), or have congenital or acquired immunodeficiency
10. Active substance abuse or a history of substance abuse within 6 months prior to Screening
11. Bacterial infections requiring treatment with oral or injectable antibiotics, or significant viral or fungal infections, within 4 weeks of Screening
12. Malignancy or history of malignancy (except for treated [ie, cured] basal cell or squamous cell in situ skin carcinomas and treated [ie, cured] cervical intraepithelial neoplasia [CIN] or carcinoma in situ of the cervix with no evidence of recurrence within the previous 5 years)
13. Psoriasis flare or rebound within 4 weeks prior to Screening
14. Evidence of skin conditions that would interfere with clinical assessments
15. Topical therapy within 2 weeks of randomization
16. Systemic therapy for psoriasis within 4 weeks prior to randomization
17. Use of phototherapy within 4 weeks prior to randomization (ie, Ultraviolet B (UVB), psoralen and ultraviolet A (PUVA)
18. Adalimumab, etanercept, infliximab, or certolizumab pegol within 12 weeks prior to randomization
19. Alefacept, briakinumab, or ustekinumab within 24 weeks prior to randomization
20. Use of any investigational drug within 4 weeks prior to randomization
21. Prolonged sun exposure or use of tanning booths or other ultraviolet (UV) light sources
22. Prior treatment with apremilast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 844 (Actual)
Dates: Start 2010-09-09 (Actual); Primary Completion 2012-02-23 (Actual); Study Completion 2016-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Reich K, Mrowietz U, Menter A, Griffiths CEM, Bagel J, Strober B, Nunez Gomez N, Shi R, Guerette B, Lebwohl M. Effect of baseline disease severity on achievement of treatment target with apremilast: results from a pooled analysis. J Eur Acad Dermatol Venereol. 2021 Dec;35(12):2409-2414. doi: 10.1111/jdv.17520. Epub 2021 Aug 23. PMID 34255891
- [Derived] Mease PJ, Hatemi G, Paris M, Cheng S, Maes P, Zhang W, Shi R, Flower A, Picard H, Stein Gold L. Apremilast Long-Term Safety Up to 5 Years from 15 Pooled Randomized, Placebo-Controlled Studies of Psoriasis, Psoriatic Arthritis, and Behcet's Syndrome. Am J Clin Dermatol. 2023 Sep;24(5):809-820. doi: 10.1007/s40257-023-00783-7. Epub 2023 Jun 14. PMID 37316690

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 76 study centers in 8 countries
Groups:
- Apremilast: Participants were initially randomized to apremilast (APR) 30 mg tablets twice daily (BID) during the Placebo-controlled Phase (Weeks 0-16)
- Placebo: Participants were initially randomized to identically matching placebo (PBO) tablets twice daily BID during the Placebo-controlled Phase (Weeks 0-16)
- Apremilast-Apremilast: Participants who were initially randomized to APR 30 mg tablets BID during the Placebo-controlled Phase (Weeks 0-16) remained on APR 30 mg BID during the Maintenance Phase (Weeks 16-32).
- Placebo-Apremilast: Participants who were initially randomized to identically matching placebo tablets BID during the Placebo-controlled Phase (Weeks 0-16) were switched after 16 weeks of treatment to apremilast 30 mg tablets BID and continued dosing with apremilast 30 mg BID during the Maintenance Phase (Weeks 16-32)
- APR-APR-Re-randomized to PBO: Participants who were initially randomized to APR 30 mg BID during the 16-week Placebo-controlled Phase (Weeks 0-16) continued dosing with APR 30 mg BID through the Maintenance Phase (Weeks 16-32). At Week 32, those participants who were considered responders [ie, having a ≥ Psoriasis Area and Severity Index score of 75 (PASI-75) response] were re-randomized to PBO during the Randomized Withdrawal Phase (Weeks 32-52). Those participants who retained their ≥PASI-75 response through the Randomized Withdrawal Phase remained on PBO until week 52. Those participants who lost their PASI-75 improvement achieved at week 32, were switched back to APR 30 mg BID at the time loss of effect was observed. All participants who completed the Randomized Withdrawal Phase at week 52 were eligible to participate in the Long-term Extension Phase from weeks 52-260, and received APR 30 mg BID for the remainder of their participation.
- APR-APR-Re-randomized to APR: Participants who were initially randomized to APR 30 mg BID during the 16-week Placebo-controlled Phase (Weeks 0-16) continued dosing with APR 30 mg BID through the Maintenance Phase (Weeks 16-32). At Week 32, those participants who were considered responders (ie, having a ≥PASI-75 response) were re-randomized to APR 30 mg BID during the Randomized Withdrawal Phase (Weeks 32-52). Those participants who completed the Randomized Withdrawal Phase at Week 52 were eligible to participate in the Long-term Extension Phase from weeks 52-260 and remained on APR 30 mg BID for the remainder of their participation.
- APR-APR-APR + Optional Topicals/UVB: Participants who were initially randomized to APR 30 mg BID during the 16-week Placebo-controlled Phase (Weeks 0-16) continued dosing with APR 30 mg BID through the Maintenance Phase (Weeks 16-32). At week 32, those participants who were considered partial responders (ie, having a response of PASI-50 to PASI-74) and non-responders (ie, having a response of <PASI-50), remained on APR 30 mg BID and were given the option of adding topical therapies and/or phototherapy to their regimen. Those participants who completed the Randomized Withdrawal Phase at week 52 were eligible to participate in the Long-term Extension Phase from weeks 52-260 and remained on APR 30 mg BID for the remainder of their participation.
- PBO-APR-APR + Optional Topicals/ UVB: Participants who were initially randomized to placebo BID during the 16-week Placebo-controlled Phase (Weeks 0-16) were switched after 16 weeks of treatment to APR 30 mg BID and continued dosing with APR 30 mg BID during the Maintenance Phase (Weeks 16-32). At week 32, all participants continued to receive APR 30mg BID. Those participants who were considered partial responders (ie, having a response of PASI-50 to PASI-74) or non-responders (ie, having a response of < PASI-50) were given the option of adding topical therapies and/or phototherapy to their regimen. A subset of these partial or non-responders received additional topical or phototherapy. All participants who completed the Randomized Withdrawal Phase at week 52 were eligible to participate in the Long-term Extension Phase from weeks 52-260 and remained on APR 30 mg BID for the remainder of their participation.
- Apremilast (Long-term Extension): Participants who were initially randomized to APR 30 mg BID during the 16-week placebo-controlled phase (Weeks 0-16) continued receiving APR 30 mg BID through the Maintenance Phase (Weeks 16-32) and were re-randomized to APR 30 mg tablets or placebo tablets BID during the Randomized Withdrawal Phase; participants were eligible to participate in the Long-term Extension Phase from Weeks 52-260 and received APR 30 mg BID for the remainder of their participation.
- Placebo-Apremilast (Long-term Extension): Participants who were initially randomized to identically matching placebo BID during the placebo-controlled phase (Weeks 0-16) were switched after 16 weeks of treatment to apremilast 30 mg tablets BID and continued dosing with apremilast 30 mg BID during the Maintenance Phase (Weeks 16-32) and Randomized Withdrawal Phase were eligible to participate in the Long-term Extension phase from Weeks 52-260 and continued on apremilast 30 mg tablets BID for the remainder of their participation.
Period: Placebo-Controlled Phase Weeks 0-16
Arm/Group | Apremilast | Placebo | Apremilast-Apremilast | Placebo-Apremilast | APR-APR-Re-randomized to PBO | APR-APR-Re-randomized to APR | APR-APR-APR + Optional Topicals/UVB | PBO-APR-APR + Optional Topicals/ UVB | Apremilast (Long-term Extension) | Placebo-Apremilast (Long-term Extension)
Started | 562 | 282 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received Apremilast | 560 | 282 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 503 | 249 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 59 | 33 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 23 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Noncompliance with study drug | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 7 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Miscellaneous | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Phase Weeks16-32
Arm/Group | Apremilast | Placebo | Apremilast-Apremilast | Placebo-Apremilast | APR-APR-Re-randomized to PBO | APR-APR-Re-randomized to APR | APR-APR-APR + Optional Topicals/UVB | PBO-APR-APR + Optional Topicals/ UVB | Apremilast (Long-term Extension) | Placebo-Apremilast (Long-term Extension)
Started | 0 | 0 | 494 (9 participants discontinued after Week 16 but prior to entry into the Maintenance Phase) | 245 (4 participants discontinued after Week 16 but prior to entry into the Maintenance Phase) | 0 | 0 | 0 | 0 | 0 | 0
Received Apremilast | 0 | 0 | 493 (1 participant elected not to participate at the time the first dose was dispensed.) | 244 (1 participant elected not to participate at the time the first dose was dispensed.) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 424 | 215 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 70 | 30 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 8 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 37 | 15 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance with Study Drug | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 12 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Randomized Withdrawal Phase-Weeks 32-52
Arm/Group | Apremilast | Placebo | Apremilast-Apremilast | Placebo-Apremilast | APR-APR-Re-randomized to PBO | APR-APR-Re-randomized to APR | APR-APR-APR + Optional Topicals/UVB | PBO-APR-APR + Optional Topicals/ UVB | Apremilast (Long-term Extension) | Placebo-Apremilast (Long-term Extension)
Started | 0 | 0 | 0 | 0 | 77 (7 participants discontinued after week 32 but prior to entry into the Randomized withdrawal Phase) | 77 (25 participants discontinued after week 32 but prior to entry into the Randomized withdrawal Phase) | 245 | 208 | 0 | 0
Received Topical + Light Therapy | 0 | 0 | 0 | 0 | 0 | 0 | 126 | 91 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 73 (1 participant discontinued after Week 52 but prior to entry into the long term extension study) | 73 (5 participants discontinued after Week 52 but prior to entry into the long term extension study) | 184 (18 participants discontinued after Week 52 but prior to entry into the long term extension study) | 163 (10 participants discontinued after Week 52 but prior to entry into the long term extension study) | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 4 | 4 | 61 | 45 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 5 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 1 | 35 | 33 | 0 | 0
Not completed — Non-compliance with Study Drug | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 12 | 6 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 2 | 5 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Long-Term Extension Weeks 52 to 260
Arm/Group | Apremilast | Placebo | Apremilast-Apremilast | Placebo-Apremilast | APR-APR-Re-randomized to PBO | APR-APR-Re-randomized to APR | APR-APR-APR + Optional Topicals/UVB | PBO-APR-APR + Optional Topicals/ UVB | Apremilast (Long-term Extension) | Placebo-Apremilast (Long-term Extension)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 306 | 153
Received at Least 1 Dose of IP | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 304 | 153
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 86 | 41
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 220 | 112
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 14
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 81 | 49
Not completed — Noncompliance with IP | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 66 | 32
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 10
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all participants who were randomized as specified in the protocol. Those who were randomized in error and did not receive any dose of Investigational product were excluded from FAS. Participants were included in the treatment group to which they were randomized APR 30 BID or placebo for the FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Apremilast | Placebo | Total
Number analyzed (Participants) | 562 | 282 | 844
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (13.07) | 46.5 (12.72) | 46.0 (12.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 88 | 271
  Male | 379 | 194 | 573
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 5 | 7
  Asian | 28 | 16 | 44
  Black or African American | 18 | 10 | 28
  Native Hawaiian or Other Pacific Islander | 5 | 1 | 6
  White | 507 | 250 | 757
  Other | 2 | 0 | 2
Duration of Plaque Psoriasis [Number; unit: years] — All participants enrolled were required to have a diagnosis of plaque psoriasis at least 12 months prior to screening, but the duration was not required for enrollment. Overall baseline population for duration of plaque psoriasis in the apremilast arm were 562 participants and 282 for those in the placebo arm.
  years
    <10 years | 150 | 85 | 235
    10 to < 20 years | 159 | 73 | 232
    ≥ 20 years | 253 | 122 | 375
    Missing | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a 75% Improvement (Response) in the Psoriasis Area Severity Index (PASI-75) at Week 16 From Baseline
Description: PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 16. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The PASI score was set to missing if any severity score or degree of involvement is missing.
Time Frame: Baseline to Week 16
Population: The Full Analysis Set (FAS) consisted of all participants who were randomized per protocol. Participants were included in the treatment group to which they were randomized APR 30 BID or placebo for the FAS. Last observation carried forward (LOCF) imputation was used.
Measure: Number; unit: percentage of participants
Groups:
- Placebo/Apremilast: Participants were initially randomized to apremilast (APR) 30 mg tablets twice daily (BID) during the Placebo-controlled Phase (Weeks 0-16)
- Placebo (PBO): Participants were initially randomized to identically matching placebo (PBO) tablets twice daily BID during the Placebo-controlled Phase (Weeks 0-16)
Arm/Group | Placebo/Apremilast | Placebo (PBO)
Number analyzed (Participants) | 562 | 282
percentage of participants | 33.1 | 5.3
Statistical Analysis 1: Comparison: Placebo/Apremilast vs Placebo (PBO); Test type: Superiority or Other; p < 0.0001, Chi-squared; Risk Difference (RD) = 27.8, 95% CI 2-sided [23.1 to 32.5]

2. Secondary Outcome: Percentage of Participants Who Achieved a Static Physician Global Assessment (sPGA) Score of Clear (0) or Almost Clear (1) With At Least 2 Points Reduction From Baseline
Description: The sPGA was a 5-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), to 4 (severe), incorporating an assessment of the severity of the three primary signs of the disease: erythema, scaling and plaque elevation. When making the assessment of overall severity, the Investigator factored in areas that have already been cleared (ie, have scores of 0) and did not just evaluate remaining lesions for severity, ie, the severity of each sign was averaged across all areas of involvement, including cleared lesions. In the event of different severities across disease signs, the sign that is the predominant feature of the disease should be used to help determine the sPGA score.
Time Frame: Baseline to Week 16
Population: The Full Analysis Set (FAS) consisted of all participants who were randomized per protocol. Participants were included in the treatment group to which they were randomized APR 30 BID or placebo for the FAS. Last observation carried forward imputation was used.
Measure: Number; unit: percentage of participants
Groups:
- Apremilast: Participants were initially randomized to apremilast 30mg tablets BID during the Placebo-controlled Phase (weeks 0-16)
- Placebo: Participants were initially randomized to identically matching placebo (PBO) tablets BID during the Placebo-controlled Phase (weeks 0-16)
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 562 | 282
percentage of participants | 21.7 | 3.9
Statistical Analysis 1: Comparison: Apremilast vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared; Risk Difference (RD) = 17.8, 95% CI 2-sided [13.7 to 21.9]

3. Secondary Outcome: Percent Change From Baseline in Percent of Affected Body Surface Area (BSA) at Week 16
Description: BSA was a measurement of involved skin. The overall BSA affected by psoriasis was estimated based on the palm area of the participant's hand (entire palmar surface or "handprint" including the fingers), which equates to approximately 1% of total body surface area. BSA percent change from baseline (Visit 2 Week 0) was determined at each visit of the study, which is calculated as 100*(visit BSA - baseline BSA) / baseline BSA (%).
Time Frame: Baseline and Week 16
Population: The Full Analysis Set (FAS) consisted of all participants who were randomized per protocol. Participants were included in the treatment group to which they were randomized APR 30 BID or placebo for the FAS. Participants with a baseline value and at least 1 postbaseline value were included. Last observation carried forward imputation was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Apremilast: Participants were initially randomized to apremilast (APR) 30 mg tablets BID during the Placebo-controlled Phase (weeks 0-16)
- Placebo: Participants were initially randomized to identically matching PBO tablets BID during the Placebo-controlled Phase (weeks 0-16)
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 559 | 278
percent change | -47.77 (1.634) [-44.56 to -50.98] | -6.99 (2.317) [-2.54 to -11.54]
Statistical Analysis 1: Comparison: Apremilast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The model included treatment group as a factor and the baseline value as a covariate. The estimation and p-value were adjusted by the covariate; Difference in LS Mean = -40.78, 95% CI 2-sided [-46.34 to -35.21]

4. Secondary Outcome: Percent Change From Baseline in the Psoriasis Area Severity Index (PASI) Score at Week 16
Description: Psoriasis Area Severity Index (PASI) scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. These values for each anatomic region are summed to yield the PASI score. The PASI score was set to missing if any severity score or degree of involvement is missing. PASI score percent change from baseline was calculated as 100* (visit score - baseline score)/baseline score (%).
Time Frame: Baseline to Week 16
Population: The Full Analysis Set (FAS) consisted of all participants who were randomized per protocol. Participants were included in the treatment group to which they were randomized APR 30 BID or placebo for the FAS. Last observation carried forward imputation was used. Participants with a baseline value and at least 1 postbaseline value are included .
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo/Apremilast | Placebo
Number analyzed (Participants) | 559 | 278
percent change | -52.1 (1.37) | -16.8 (1.94)
Statistical Analysis 1: Comparison: Placebo/Apremilast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 3, analysis 1]; Difference in LS Mean = -35.3, 95% CI 2-sided [-39.9 to -30.6]

5. Secondary Outcome: Percentage of Participants Who Achieved a 50% Improvement (Response) in the PASI Score (PASI-50) at Week 16 From Baseline
Description: A participant was classified as having at least a 50% improvement in PASI score from baseline, which was equivalent to a percent change from baseline ranging from -100% to -50%. PASI score is based on an assessment of erythema (reddening), induration (plaque thickness), desquamation (scaling), and the percent area affected as observed on the day of examination.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo/Apremilast | Placebo
Number analyzed (Participants) | 562 | 282
Percentage of Participants | 58.7 | 17.0
Statistical Analysis 1: Comparison: Placebo/Apremilast vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared; Risk Difference (RD) = 41.7, 95% CI 2-sided [35.7 to 47.7]

6. Secondary Outcome: Change From Baseline in Pruritus Visual Analog Scale (VAS) Score at Week 16
Description: The Pruritus Visual Analog Scores (VAS) were used to measure the amount of itching and discomfort a participant experiences. Participant's Assessment of Pruritus (Itch) asked: On average, how much itch have you had because of your condition in the past week? All VAS values range from 0 to 100. Higher scores correspond to more severe symptom or disease. Change from baseline was calculated for the VAS scale, where change = visit value - baseline value.
Time Frame: Baseline and Week 16
Population: The Full Analysis Set (FAS) consisted of all participants who were randomized per protocol. Participants were included in the treatment group to which they were randomized APR 30 BID or placebo for the FAS. Last observation carried forward imputation was used. Participants with a baseline value and at least 1 postbaseline value are included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 559 | 277
units on a scale | -31.5 (1.30) | -7.3 (1.85)
Statistical Analysis 1: Comparison: Apremilast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA; Based on an analysis of variance model for the change from baseline at Week 16, with treatment group as a factor (an ANOVA model); Difference in LS Mean = -24.2, 95% CI 2-sided [-28.7 to -19.8]

7. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI) Total Score at Week 16
Description: DLQI is a simple, compact, and practical questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. With the exception of Item Number 7, the participant responds on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). Item Number 7 is a multi-part item, the first part of which ascertains whether the participant's skin prevented them from working or studying (Yes or No, scores 3 or 0 respectively), and if "No," then the participant is asked how much of a problem the skin has been at work or study over the past week, with response alternatives being "A lot," "A little," or "Not at all" (scores 2, 1, or 0 respectively). The DLQI total score is derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best.
Time Frame: Baseline to Week 16
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 556 | 274
units on a scale | -6.6 (0.27) | -2.1 (0.38)
Statistical Analysis 1: Comparison: Apremilast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA; Difference in LS Mean = -4.5, 95% CI 2-sided [-5.4 to -3.6] — Based on an analysis of covariance model for the change from baseline at Week 16, with treatment group as a factor, the baseline value, and the treatment by baseline interaction term as covariates

8. Secondary Outcome: Change From Baseline in the Mental Component Summary (MSC) Score of the Medical Outcome Study Short Form 36-item (SF-36) Health Survey Version 2.0 at Week 16
Description: The SF-36 was a 36-item general health status instrument and consists of 8 scales: physical function (PF), role limitations-physical (RP), vitality (VT), general health perceptions (GH), bodily pain (BP), social function (SF), role limitations-emotional (RE), and mental health (MH). Scale scores range from 0 to 100, with higher scores indicating better health. Two overall summary scores were obtained - a Physical Component Summary score (PCS) and a Mental Component Summary score (MCS). Scores from the 8 scales, PCS and MCS were transformed to the norm-based scores using weights from U.S. general population, with 50 as the average and 10 as the standard deviation, higher scores indicating better health. For norm based scores, change from baseline were calculated for the 8 scales and the two summary scales, where change = visit value - baseline value.
Time Frame: Baseline to Week 16
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 556 | 273
units on a scale | 2.28 (0.371) | -0.81 (0.529)
Statistical Analysis 1: Comparison: Apremilast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = 3.08, 95% CI 2-sided [1.81 to 4.35]

9. Secondary Outcome: Percentage of Participants Who Achieved Both a 75% Improvement (Response) in the PASI and sPGA Score of Clear (0) or Almost Clear (1) With at Least 2 Points Reduction at Week 16 From Baseline
Description: PASI-75 response was the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 16. The improvement in PASI score was used as a measure of efficacy. See Outcome Measure #1 for further description. sPGA is a 5-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), to 4 (severe), incorporating an assessment of the severity of the three primary signs of the disease: erythema, scaling and plaque elevation. See OCM #2 for further description.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 562 | 282
percentage of participants | 20.3 | 3.5
Statistical Analysis 1: Comparison: Apremilast vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared; Risk Difference (RD) = 16.7, 95% CI 2-sided [12.8 to 20.7]

10. Secondary Outcome: Kaplan Meier Estimate of Time to Loss of PASI-75 Response (Loss of Effect) at Week 32 During the Re-Randomized Treatment Withdrawal Phase
Description: Time to loss was the time between the re-randomization date and the date of the first assessment where loss of PASI-75 was observed (event); or the time between the re-randomization date and the date of the last PASI assessment in the Weeks 32-52 interval prior to addition of protocol-prohibited medication/therapy, or resumption of APR 30 BID, or discontinuation, or Week 52 if no loss (censored).
Time Frame: Week 32 to Week 52
Population: Analysis population consisted of participants who were re-randomized to placebo or apremilast 30mg BID at Week 32.
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- APR-APR -Re-randomized to PBO: Participants who were initially randomized to APR 30 mg BID during the 16-week Placebo-controlled Phase continued dosing with APR 30 mg BID through the Maintenance Phase (weeks 16-32). At Week 32, those participants who were considered responders (ie, having a ≥PASI-75 response) were re-randomized to PBO during the Randomized Withdrawal Phase (Weeks 32-52). Those participants who retained their ≥PASI-75 response through the Randomized Withdrawal Phase remained on PBO until Week 52. Those participants who lost their PASI-75 improvement achieved at Week 32, were switched back to APR 30 mg BID at the time loss of effect was observed.
Arm/Group | APR-APR-Re-randomized to APR | APR-APR -Re-randomized to PBO
Number analyzed (Participants) | 77 | 77
Weeks | 17.7 [13.0 to NA] — The upper limit was not available since there were not enough participants who lost response by the end of the Randomized Withdrawal Phase for the estimation. | 5.1 [4.1 to 8.1]
Statistical Analysis 1: Comparison: APR-APR-Re-randomized to APR vs APR-APR -Re-randomized to PBO; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 2.649, 95% CI 2-sided [1.768 to 3.969]

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) During the Placebo-Controlled Phase
Description: An AE was any noxious, unintended, or untoward medical occurrence, that may appear or worsen in a participant during the course of study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) was considered an AE. A serious AE (SAE) is any untoward adverse event that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly or birth defect, or a condition that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above. An AE is a treatment emergent AE if the AE start date is on or after the date of the first dose of study drug and no later than 28 days after the last dose.
Time Frame: Week 0 to Week 16; mean duration of exposure was 14.8 weeks and 15.0 weeks for subjects randomized to placebo and apremilast respectively.
Population: Safety population consisted of all participants who were randomized and received at least one dose of Investigational Product (IP)
Measure: Number; unit: participants
Groups:
- Apremilast: Participants were initially randomized to apremilast 30 mg tablets BID during the Placebo-controlled Phase (weeks 0-16)
- Placebo: Participants were initially randomized to identically matching placebo tablets BID during the Placebo-controlled Phase (weeks 0-16)
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 560 | 282
participants
  Any TEAE | 388 | 157
  Any Drug-Related TEAE | 224 | 58
  Any Severe TEAE | 20 | 9
  Any Serious TEAE | 12 | 8
  Any Serious Drug-Related TEAE | 4 | 0
  Any TEAE leading to Drug Interruption | 37 | 13
  Any TEAE leading to drug withdrawal | 29 | 9
  Any TEAE Leading to Death | 1 | 1

12. Secondary Outcome: Number of Participants With TEAEs During the Apremilast-Exposure Period Through Week 260
Description: The Apremilast-exposure Period started on the date of the first dose of apremilast (Week 0 for participants originally randomized to apremilast or Week 16 for participants originally randomized to placebo) to the last dose of apremilast. Adverse events that started after 28 days of initiating placebo and before resuming apremilast treatment in the Randomized Treatment Withdrawal Phase (Weeks 32 to 52) were excluded in the Apremilast-exposure Period. A serious AE (SAE) is any untoward adverse event that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly or birth defect, or a condition that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above. An AE is a treatment emergent AE if the AE start date is on or after the date of the first dose of study drug and no later than 28 days after the last dose.
Time Frame: Week 0 to Week 260; mean exposure to apremilast 30 mg BID during the Apremilast-exposure Period up to Week 260 was 97.83 weeks
Population: The apremilast subjects as treated population, which includes all participants who were randomized to (at Week 0) or treated with (at Week 16) apremilast 30 mg BID, and received at least one dose of apremilast after randomization or Week 16.
Measure: Number; unit: participants
Groups:
- Apremilast: Participants initially randomized to placebo or apremilast 30 mg tablets BID during the 16-week placebo-controlled phase (Weeks 0-16) continued to receive apremilast 30 mg BID through the maintenance phase; during the randomized withdrawal phase (Weeks 32-52) participants continued to receive apremilast 30 mg BID or were again randomized to either apremilast 30 mg BID or placebo and were transitioned to apremilast 30 mg BID after loss of response or in the long-term extension phase from Weeks 52-260,
Arm/Group | Apremilast
Number analyzed (Participants) | 804
participants
  Any At TEAE | 675
  Any Drug-Related TEAE | 372
  Any Severe TEAE | 78
  Any Serious TEAE | 74
  Any Serious Drug-Related TEAE | 12
  Any TEAE Leading to Drug Interruption | 107
  Any TEAE Leading to Drug withdrawal | 98
  Any TEAE Leading to Death | 3

13. Secondary Outcome: Number of Participants With a Psoriasis Flare or Rebound During the Placebo-Controlled Phase
Description: Psoriasis flare was defined as a sudden intensification of psoriasis requiring medical intervention, or a diagnosis of new generalized erythrodermic, inflammatory, or pustular psoriasis. Rebound is defined as a severe and sudden worsening of disease that occurs after treatment has been discontinued. Note categories below. [1] Psoriasis adverse events (ie, preferred term as Guttate psoriasis, Psoriasis, Pustular psoriasis) started on or after the first dose date and on or before the last dose date within the phase. [2] Psoriasis adverse events (ie, preferred term as Guttate psoriasis, Psoriasis, Pustular psoriasis, Rebound psoriasis) started after the last dose date for participants who discontinued within the phase. [3] PASI >= 125% of baseline score at any visit after the last dose date for participants who discontinued within the phase and were not included in [1] and/or [2].
Time Frame: Weeks 0 to Week 16
Population: Included all participants who were randomized and received at least one dose of Investigational Product (IP).
Measure: Number; unit: participants
Groups:
- Placebo: Participants were initially randomized to placebo tablets BID during the Placebo-controlled Phase (Weeks 0-16)
Arm/Group | Placebo | Apremilast
Number analyzed (Participants) | 282 | 560
participants
  Participants with any psoriasis flare [1] | 7 | 6
  Participants with any psoriasis rebound [2] | 1 | 1
  PASI ≥ 125% of Baseline score after last dose [3] | 3 | 3

14. Secondary Outcome: Number of Participants With a Psoriasis Flare or Rebound During the During the Apremilast-exposure Period Through Week 260
Description: as for outcome 13
Time Frame: Week 0 to Week 260
Population: Safety population consisted of all participants who were randomized and received at least one dose of IP; apremilast participants as treated
Measure: Number; unit: participants
Groups:
- Apremilast: Participants initially randomized to placebo or apremilast 30 mg tablets BID during the 16-week placebo-controlled phase (Weeks 0-16) continued to receive apremilast 30 mg BID through the maintenance phase; during the randomized withdrawal phase (Weeks 32-52) participants continued to receive apremilast 30 mg BID or were again randomized to either apremilast 30 mg BID or placebo and were transitioned to apremilast 30 mg BID after loss of response or in the long-term extension phase from Weeks 52-260
Arm/Group | Apremilast
Number analyzed (Participants) | 804
participants
  Participants with any psoriasis flare [1] | 35
  Participants with any psoriasis rebound [2] | 12
  PASI ≥ 125% of Baseline score after last dose [3] | 26

ADVERSE EVENTS:
Time Frame: AEs are reported at: 1. Weeks 0-16: PBO-controlled phase 2. Weeks 32-52 Randomized Withdrawal participants re-randomized to PBO at Week 32 3. Weeks 0-260 APR-exposure period for participants randomized or switched to APR at any time during the study
Description: During the PBO-controlled Phase (Weeks 0-16), the mean duration of treatment for those randomized to APR 30 BID or PBO at Week 0, was 15.0 and 14.8, respectively; for those re-randomized to PBO at Week 32, the mean duration of PBO was 8.1 weeks; during the APR-Exposure Period (Weeks 0-260), the mean duration of exposure to APR was 97.83 weeks
Groups:
- Placebo (Placebo-Controlled Phase) Weeks 0-16: Participants randomized and received identically matching placebo tablets BID during the Placebo-controlled Phase (Weeks 0-16)
- Apremilast (Placebo-Controlled Phase) Weeks 0-16: Participants randomized and received apremilast 30 mg tablets BID during the Placebo-Controlled Phase (Weeks 0-16)
- APR-APR-PBO Randomized Withdrawal Phase Weeks 32-52: Participants re-randomized and received placebo tablets BID at Week 32. Data from Week 32 up to Week 52 when participants received placebo treatment.
- Apremilast (Apremilast Exposure Period) Weeks 0-260: Participants who received apremilast 30 mg tablets BID, regardless of when the apremilast exposure started (at Week 0 or at week 16), up until Week 260. Adverse events associated with apremilast treatment up to Week 260 were included. AEs that started more than 28 days after Placebo treatment and prior to resuming apremilast were excluded for participants who were re-randomized to Placebo at Week 32.
Arm/Group | Placebo (Placebo-Controlled Phase) Weeks 0-16 | Apremilast (Placebo-Controlled Phase) Weeks 0-16 | APR-APR-PBO Randomized Withdrawal Phase Weeks 32-52 | Apremilast (Apremilast Exposure Period) Weeks 0-260
Serious Adverse Events (participants affected / at risk) | 8/282 | 12/560 | 2/77 | 74/804
Other Adverse Events (participants affected / at risk) | 90/282 | 260/560 | 10/77 | 503/804
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Placebo-Controlled Phase) Weeks 0-16 (N=282) | Apremilast (Placebo-Controlled Phase) Weeks 0-16 (N=560) | APR-APR-PBO Randomized Withdrawal Phase Weeks 32-52 (N=77) | Apremilast (Apremilast Exposure Period) Weeks 0-260 (N=804)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 4
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 6
Mitral valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Leukoplakia oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 2
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Chemical burns of eye (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Conjunctival primary acquired melanosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 2
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 4
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Placebo-Controlled Phase) Weeks 0-16 (N=282) | Apremilast (Placebo-Controlled Phase) Weeks 0-16 (N=560) | APR-APR-PBO Randomized Withdrawal Phase Weeks 32-52 (N=77) | Apremilast (Apremilast Exposure Period) Weeks 0-260 (N=804)
Diarrhoea (Gastrointestinal disorders) | 20 | 105 | 0 | 163
Nausea (Gastrointestinal disorders) | 19 | 88 | 0 | 130
Gastroenteritis (Infections and infestations) | 6 | 10 | 0 | 41
Nasopharyngitis (Infections and infestations) | 23 | 41 | 3 | 131
Sinusitis (Infections and infestations) | 5 | 16 | 1 | 45
Upper respiratory tract infection (Infections and infestations) | 21 | 57 | 2 | 183
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 9 | 2 | 51
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 14 | 1 | 50
Headache (Nervous system disorders) | 13 | 31 | 0 | 62
Tension headache (Nervous system disorders) | 12 | 41 | 2 | 84
Hypertension (Vascular disorders) | 7 | 10 | 0 | 56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.